CLINICAL TRIAL: NCT03287102
Title: Dissociated Optic Nerve Fiber Layer Appearance and Retinal Sensitivity After Macular Hole Surgery With Temporal Inverted Internal Limiting Membrane Flap Technique
Brief Title: Macular Hole Surgery With Temporal Inverted Internal Limiting Membrane Flap (MARTIAL)
Acronym: MARTIAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-A02061-52
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-09

CONDITIONS: Macula Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporal inverted ILM peeling group (Other): The internal limiting membrane is peeled from the temporal side of the fovea only
  Interventions: Procedure: Macular hole surgery
- Complete ILM peeling group (Other): The internal limiting membrane is completely removed around the fovea
  Interventions: Procedure: Macular hole surgery

INTERVENTIONS:
Procedure: Macular hole surgery — Vitrectomy, temporal inverted or complete ILM peeling and gas tamponade

SUMMARY:
Since 1991, idiopathic macular holes (MH) can benefit from an effective treatment initially involving pars plana vitrectomy, stripping of epiretinal membranes and intraocular gas tamponade followed by facedown positioning. The initial 58% success rate has further increased to 85-100% with internal limiting membrane (ILM) peeling. However, complete ILM removal has been shown to lead to anatomic changes causing the retina to have the appearance of a dissociated optic nerve fiber layer (DONFL). Moreover, it has been associated with decreased retinal sensitivity that may cause visual discomfort despite good visual acuity. Nawrocki et al. recently suggested to reduce the area of peeled ILM (temporal inverted ILM flap technique) in order to minimize iatrogenic trauma while maintaining satisfactory surgical outcomes. The aim of this study is to compare the incidence of DONFL appearance and retinal sensitivity after macular hole surgery in eyes that underwent temporal inverted ILM flap technique and eyes that had complete ILM peeling

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old

Exclusion Criteria:

* Underage patients
* History of intraocular surgery (except for cataract surgery)
* Macular hole secondary to trauma, diabetic retinopathy, uveitis or associated with retinal detachment
* Concurrent macular disease (diabetic maculopathy, age-related macular degeneration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of dimples on optical coherence tomography | 3 months after surgery
  Incidence of DONFL appearance

SECONDARY OUTCOMES:
Retinal sensitivity on microperimetry testing (decibel) | 3 months after surgery
Macular hole closure rate on optical coherence tomography | 3 months after surgery
Visual acuity (Logarithm of the Minimum Angle of Resolution) | 3 months after surgery
Ellipsoide zone defect on optical coherence tomography | 3 months after surgery
External limiting membrane defect on optical coherence tomography | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste CONART, Principal Investigator — Brabois Hospital, Nancy, France
Locations (1):
- Brabois Hospital, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michalewska Z, Michalewski J, Dulczewska-Cichecka K, Adelman RA, Nawrocki J. TEMPORAL INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE VERSUS CLASSIC INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE: A Comparative Study. Retina. 2015 Sep;35(9):1844-50. doi: 10.1097/IAE.0000000000000555. PMID 25946691
- [Background] Michalewska Z, Michalewski J, Dulczewska-Cichecka K, Nawrocki J. Inverted internal limiting membrane flap technique for surgical repair of myopic macular holes. Retina. 2014 Apr;34(4):664-9. doi: 10.1097/IAE.0000000000000042. PMID 24263468
- [Background] Tadayoni R, Svorenova I, Erginay A, Gaudric A, Massin P. Decreased retinal sensitivity after internal limiting membrane peeling for macular hole surgery. Br J Ophthalmol. 2012 Dec;96(12):1513-6. doi: 10.1136/bjophthalmol-2012-302035. Epub 2012 Oct 17. PMID 23077227
- [Background] Michalewska Z, Michalewski J, Adelman RA, Nawrocki J. Inverted internal limiting membrane flap technique for large macular holes. Ophthalmology. 2010 Oct;117(10):2018-25. doi: 10.1016/j.ophtha.2010.02.011. Epub 2010 Jun 11. PMID 20541263
- [Background] Tadayoni R, Paques M, Massin P, Mouki-Benani S, Mikol J, Gaudric A. Dissociated optic nerve fiber layer appearance of the fundus after idiopathic epiretinal membrane removal. Ophthalmology. 2001 Dec;108(12):2279-83. doi: 10.1016/s0161-6420(01)00856-9. PMID 11733271